CLINICAL TRIAL: NCT05776849
Title: The Effect of Flipped Classroom Design on Episiotomy Teaching on Knowledge, Skills and Anxiety Levels of Midwifery Students: A Randomized Controlled Study
Brief Title: Flipped Classroom in Episiotomy Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, yasemin hamlacı başkaya, Head of Midwifery Depatment, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 01032023
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Flipped Classroom; Episiotomy
Keywords: Flipped classroom; midwifery; episiotomy; anxiety; student
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: the experimental group will be given the teaching materials before the lesson, while the control group will be given them during the lesson
Who Masked: Outcomes Assessor
Masking Description: The person assessing the outcomes was blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The trainer shared the training presentation, visuals and videos (his own video explaining the episiotomy application and repair and other videos shared with the traditional group) prepared on the subject of episiotomy with the students through the course information system, one week before the episiotomy application. It was accepted that the students came to the episiotomy application with the theoretical training. Afterwards, episiotomy was applied.
  Interventions: Other: flipped classroom
- No Intervention: Control group (Traditional education) (No Intervention): The students were given theoretical training. This training was implemented in two sessions, one lasting 50 minutes and the other 30 minutes. The content of the training; It included the definition of episiotomy, indications, risks, episiotomy application steps, materials used, episiotomy types, episiotomy repair and repair steps, suturing techniques and types, episiotomy care. Slide shows, related images and video presentations (3 videos showing episiotomy application and repair steps and suturing techniques) were used as teaching materials. A question-answer session was held at the end of the training. In addition, teaching materials were shared with the students after the application. Immediately after the training, episiotomy was applied.

INTERVENTIONS:
Other: flipped classroom — Educational presentation, visuals and videos (her own video explaining episiotomy application and repair and other videos shared with the traditional group) prepared for the students on episiotomy were shared one week before the episiotomy application.
  Arms: Experimental group

SUMMARY:
This study aims to evaluate the effect of using inverted classroom design on students' knowledge, skills and anxiety levels in teaching episiotomy application and repair, one of the interventions frequently used in labour.

DETAILED DESCRIPTION:
The flipped classroom is a new and popular teaching model in which lessons traditionally conducted in the classroom become homework or homework responsibilities and lessons that would normally constitute homework become classroom lessons. In the flipped classroom, students become responsible for their own learning process and need to manage their own pace of learning, while the teacher helps the students instead of simply imparting information. While flipped classrooms are seen to offer many positive educational outcomes, they also have some limitations. In the flipped model, student learning achievement and satisfaction can be increased and it is considered to be more economical than traditional teaching. The literature shows that the flipped teaching model requires both opportunities and challenges. Within the scope of the study, in order to evaluate the effect of using inverted classroom design in teaching episiotomy application and repair on students' knowledge, skills and anxiety levels, midwifery students taking normal birth and postnatal period courses will be divided into two groups, one group in the form of traditional teaching and one group in the form of inverted classroom design during the application of episiotomy teaching. The study data will be collected through Student Identification Form, State Anxiety Inventory, Episiotomy Information Form and Episiotomy Skill Evaluation Form. The data obtained from the study will be analysed with SPSS programme. It is thought that the study will make an important contribution to the literature in terms of evaluating the effect of the inverted classroom on teaching episiotomy repair.

ELIGIBILITY:
Inclusion Criteria:

1. Registered in the midwifery department,
2. Participating in the Normal Birth and Postpartum Period course during the study period and
3. Those who agreed to participate in the study

Exclusion Criteria:

1. Those who do not attend the Normal Birth and Postpartum Term course twice or more during the semester,
2. Those who have taken this course before and have experience in episiotomy skills.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
State Anxiety Inventory (STAI) | 1 hours
  The State Anxiety Inventory consists of 20 items and requires the individual to answer how he or she feels at a certain moment and under certain conditions, taking into account his feelings about the situation he is in. The scale is likert type and is a four-degree scale ranging from "Not at all" to "Totally". The maximum score that can be obtained from the scale is 80, and the minimum score is 20. High scores indicate high anxiety, low scores indicate low anxiety.
Episiotomy Information Form | 1 hours
  It consists of 25 propositions (questions) to measure the knowledge level of students about episiotomy. 13 of these propositions were prepared as true propositions and 12 as false propositions, and the participants were asked to answer as 'agree', 'disagree' and 'no idea'. Correct answers given by the students to the propositions were evaluated as 1 point, wrong and I have no idea answers as 0 points. The lowest score that can be obtained from the information form is 0, and the highest score is 25.
Episiotomy Skill Assessment Form | 1 hours
  Form; It consists of 15 items, including the steps of holding the porthole correctly, knotting the sutures properly, repairing the superficial perineal muscles with one-by-one sutures, and application and repair of episiotomy. Each item in the form was scored as "3" if the student fulfilled the procedure in the item, "2" if partially fulfilled, and "1" if not. The total score that can be obtained from the form is minimum 15 and maximum 75.

CONTACTS AND LOCATIONS:
Overall Officials: yasemin hamlacı başkaya, Study Director — Sakarya University
Locations (1):
- Sakarya University- Faculty of Health Sciences, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rotellar C, Cain J. Research, Perspectives, and Recommendations on Implementing the Flipped Classroom. Am J Pharm Educ. 2016 Mar 25;80(2):34. doi: 10.5688/ajpe80234. PMID 27073287
- [Background] Smith KM, Geletta S, Duelfer K. Flipped Classroom in Podiatric Medical Education. J Am Podiatr Med Assoc. 2020 Sep 1;110(5):Article_11. doi: 10.7547/19-060. PMID 33179058
- [Background] Youhasan P, Chen Y, Lyndon M, Henning MA. Exploring the pedagogical design features of the flipped classroom in undergraduate nursing education: a systematic review. BMC Nurs. 2021 Mar 22;20(1):50. doi: 10.1186/s12912-021-00555-w. PMID 33752654
- [Background] Vanka A, Vanka S, Wali O. Flipped classroom in dental education: A scoping review. Eur J Dent Educ. 2020 May;24(2):213-226. doi: 10.1111/eje.12487. Epub 2019 Dec 18. PMID 31808231
- [Background] Golaki SP, Kamali F, Bagherzadeh R, Hajinejad F, Vahedparast H. The effect of Flipped Classroom through Near Peer Education (FC through NPE) on patient safety knowledge retention in nursing and midwifery students: a solomon four-group design. BMC Med Educ. 2022 Feb 19;22(1):112. doi: 10.1186/s12909-022-03144-w. PMID 35183160
- [Background] Aksoy B, Pasli Gurdogan E. Examining effects of the flipped classroom approach on motivation, learning strategies, urinary system knowledge, and urinary catheterization skills of first-year nursing students. Jpn J Nurs Sci. 2022 Apr;19(2):e12469. doi: 10.1111/jjns.12469. Epub 2022 Jan 4. PMID 34984830
- [Background] Clesse C, Lighezzolo-Alnot J, De Lavergne S, Hamlin S, Scheffler M. Factors related to episiotomy practice: an evidence-based medicine systematic review. J Obstet Gynaecol. 2019 Aug;39(6):737-747. doi: 10.1080/01443615.2019.1581741. Epub 2019 Apr 25. PMID 31020867